CLINICAL TRIAL: NCT05266534
Title: The Effect of Intramyometrial Injection of Terlipressin Versus Carbitocin on Hemoglobin and Blood Loss During Open Myomectomy Operations Without Using Haemostatic Tourniquets.
Acronym: myomectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wael Elbanna Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Elbanna_008
Record Dates: First submitted 2021-12-21; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2021-12

CONDITIONS: Myoma
MeSH Terms: conditions — Myoma | interventions — Terlipressin; carbetocin; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Double Blinded Randomized Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double Blinded Randomized Placebo-Controlled Trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intramyometrial Terlipressin injection in women undergoing open myomectomy (Active Comparator): intramyometrial Terlipressin injection
  Interventions: Drug: Terlipressin
- intramyometrial Carbetocin injection in women undergoing open myomectomy (Active Comparator): intramyometrial Carbetocin injection
  Interventions: Drug: Carbetocin
- intramyometrial saline injection in women undergoing open myomectomy procedure (Placebo Comparator): intramyometrial saline injection in women
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Terlipressin — the efficacy of intramyometrial Terlipressin injection on hemoglobin level and decreasing blood loss in women undergoing open myomectomy
  Other Names: glypressin
  Arms: intramyometrial Terlipressin injection in women undergoing open myomectomy
Drug: Carbetocin — the efficacy of intramyometrial carbetocin injection on hemoglobin level and decreasing blood loss in women undergoing open myomectomy
  Other Names: pabal
  Arms: intramyometrial Carbetocin injection in women undergoing open myomectomy
Drug: Saline — the efficacy of intramyometrial saline injection on hemoglobin level and decreasing blood loss in women undergoing open myomectomy
  Other Names: NaCl 0.9
  Arms: intramyometrial saline injection in women undergoing open myomectomy procedure

SUMMARY:
For gynecologists, reaching a conclusion about the efficacy of intramyometrial Terlipressin injection versus intramyometrial Carbetocin injection on hemoglobin level and decreasing blood loss in women undergoing open myomectomy that would influence the clinical decision and best practice. Besides enriching the clinical evidence in open myomectomy without using haemostatic tourniquets. For society, our conclusion and recommendation shall maximize the benefits and managing the benefits of the technique used. Moreover, providing more information for women undergoing open myomectomy without using haemostatic tourniquets.

DETAILED DESCRIPTION:
This study is a prospective, comparative, double-blinded randomized placebo-controlled trial and multi-center study that will be conducted at Wael ElBanna Clinic and the NRC site. The study participants' relevant medical records will be collected and reviewed after obtaining informed consent for the participants. Data will be pooled and presented in aggregate, without the identification of individual subjects. The study materials that will be used will include blood tests and ultrasound. The study will involve three study arms:

* Arm 1: intramyometrial Terlipressin injection in women undergoing open myomectomy procedure without using haemostatic tourniquets
* Arm 2: intramyometrial Carbetocin injection in women undergoing open myomectomy procedure without using haemostatic tourniquets
* Arm 3: intramyometrial saline injection in women undergoing open myomectomy procedure without using haemostatic tourniquets Subjects who meet diagnostic requirements as listed in the inclusion and exclusion criteria will be included in the study. Women will be randomized to one of the three arms using a computergenerated randomization table with a 1:1:1 group allocation

ELIGIBILITY:
Inclusion Criteri

* Women aged 16-45 yearsAppropriate medical status for open surgery (Largest Myoma size from 4 cm up to 20 cm)
* Baseline hemoglobin ≥9 g/dl
* No contra-indications to the use of glyopressin or carbitocin
* Myoma-related symptoms, such as pelvic pressure or pain,menorrhagia, or infertility
* Not pregnant at the time of presentation (i.e., negative urine pregnancy test or last menstrual period within the last 4 weeks)

Exclusion Criteria

* Open myomectomy using mechanical tourniquet
* Previous myomectomy
* History of bleeding disorders
* Concurrent anticoagulation therapy
* History of Uncontrolled ischaemic heart disease
* Any pelvic abnormalities requiring concomitant surgery
* Treatment with a GnRH agonist or ulipristal acetate within three months preceding surgery
* Inability to understand and provide written informed consent

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — women with utrine fibroids
Enrollment: 162 (Estimated)
Dates: Start 2021-12-30 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
To measure the volume of intraoperative blood loss in each group without using haemostatic tourniquets | 12 hours
  the volume of intraoperative blood loss in ml myomectomy without using haemostatic tourniquets

SECONDARY OUTCOMES:
To measure the pre and postoperative hemoglobin level without using haemostatic tourniquets | 24 hours
  To measure the pre and postoperative hemoglobin level without using haemostatic tourniquets
To measure the operative time in each group without using haemostatic tourniquets | 24 hours
  To measure the operative time in each group without using haemostatic tourniquets
to assess the measure the severity of pain using VAS score | 24 hours
  post operative pain VAS score

CONTACTS AND LOCATIONS:
Locations (1):
- Wael El Banna Clinic, Maadi, Egypt

REFERENCES:
- [Background] Parker WH, Berek JS, Pritts EA, Olive D, Chalas E, Clarke-Pearson D. Regarding "Incidence of Occult Uterine Malignancy Following Vaginal Hysterectomy with Morcellation". J Minim Invasive Gynecol. 2018 Jan;25(1):187-188. doi: 10.1016/j.jmig.2017.07.027. Epub 2017 Aug 18. No abstract available. PMID 28826956
- See also: Related Info — https://www.uchicagomedicine.org/conditions-services/obgyn/uterine-fibroids?_vsrefdom=fibriods_google&gclid=EAIaIQobChMIoNvX8Zr19AIVI49oCR3CpgjaEAAYASAAEgLLn_D_BwE